CLINICAL TRIAL: NCT01474200
Title: Aquapheresis Versus Intravenous Diuretics and Hospitalizations for Heart Failure (AVOID-HF)
Brief Title: Study of Heart Failure Hospitalizations After Aquapheresis Therapy Compared to Intravenous (IV) Diuretic Treatment
Acronym: AVOID-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed due to patient recruitment challenges. No interim analyses were completed; study closure was not related to any concerns about safety or futility.
Sponsor: Nuwellis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1494
Record Dates: First submitted 2011-11-11; First posted 2011-11-18 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure; Cardiac Failure; Acute Decompensated Heart Failure (ADHF)
Keywords: Ultrafiltration; Aquapheresis; Diuretics; Loop Diuretics; Aquadex Flexflow System; Gambro UF Solutions
MeSH Terms: conditions — Heart Failure | interventions — Ultrafiltration; Sodium Potassium Chloride Symporter Inhibitors; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aquapheresis (AQ) - isolated veno-venous ultrafiltration (Experimental): Excess fluid from the patient is removed by isolated veno-venous ultrafiltration treatment using the Aquadex Flex Flow System
  Interventions: Device: Isolated veno-venous ultrafiltration (AQ)
- IV Loop Diuretics (LD) (Active Comparator): Excess fluid from the patient is removed by IV (Intravenous) loop diuretic treatment
  Interventions: Drug: IV Loop Diuretics (LD)

INTERVENTIONS:
Device: Isolated veno-venous ultrafiltration (AQ) — Aquapheresis treatment (isolated veno-venous ultrafiltration) using the Aquadex FlexFlow System during index hospitalization until the patient's signs and symptoms of fluid overload have improved to the satisfaction of the treating physician. Ultrafiltration rates, duration and frequency of treatment are dependent on the amount of patient fluid excess and on the rate of fluid movement from the interstitial spaces into the vascular compartment during Aquapheresis (Plasma Refill Rate, or PRR)
  Other Names: Aquapheresis; Ultrafiltration; Aquadex FlexFlow System; Gambro UF Solutions
  Arms: Aquapheresis (AQ) - isolated veno-venous ultrafiltration
Drug: IV Loop Diuretics (LD) — IV Loop Diuretics treatment using only FDA approved IV loop diuretics indicated for the treatment of patients with fluid overload. This includes furosemide or other IV loop diuretics administered at equivalent doses to furosemide. Patients will receive either a twice daily IV bolus or continuous IV LD infusions according to the high dose protocol of the"Diuretic strategies in patients wth acute decompensated heart failure" (DOSE) trial.
  Other Names: furosemide
  Arms: IV Loop Diuretics (LD)

SUMMARY:
The purpose of the research is to determine if patients have fewer Heart Failure (HF) events after receiving Aquapheresis (AQ) therapy compared to intravenous (IV) diuretics up to 90 days of discharge from the hospital. Heart Failure events are defined as returning to the hospital, clinic or emergency department (ED) for treatment of HF symptoms.

DETAILED DESCRIPTION:
The aim of the proposed AVOID-HF study is to confirm and expand the findings that fluid removal by AQ reduces HF rehospitalizations at 90 days as well as the length of these HF rehospitalizations. In the "Ultrafiltration Versus Intravenous Diuretics for Patients Hospitalized for Acute Decompensated Heart Failure" (UNLOAD) study, the 90 day HF re-hospitalizations were pre-specified secondary end-points. AVOID-HF is designed with a primary end-point to determine if AQ reduces the number of HF events (Rehospitalization or unscheduled outpatient or emergency room treatment for HF) after discharge from index hospitalization compared to IV loop diuretics. AVOID will also explore days alive and out of the hospital as a secondary end-point, which was not done in UNLOAD. In other words, the AVOID-HF study is going beyond studying only the amount of fluid removal and will explore whether the modality of fluid removal influences HF outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Male or non-pregnant female patients
3. Admitted to the hospital with a primary diagnosis of acute decompensated heart failure (ADHF)
4. On regularly scheduled oral loop diuretics prior to admission
5. Fluid overload manifested by at least two of the following:

   1. Pitting edema (2+) of the lower extremities
   2. Jugular venous distention > 8 cm
   3. Pulmonary edema or pleural effusion on chest x-ray
   4. Paroxysmal nocturnal dyspnea or ≥ two- pillow orthopnea
   5. Respiration rate ≥ 20 per minute.
6. Have received ≤ 2 IV loop diuretics doses before randomization
7. Must be able to be enrolled into the trial ≤ 24 hours of their admission to the hospital.
8. Provide written informed consent form as required by the local IRB (Institutional Review Board)

Exclusion Criteria:

1. Acute coronary syndromes
2. Renal insufficiency with a sCr ≥ 3.0 mg/dl or planned renal replacement therapies
3. Systolic blood pressure < 90 mmHg at time of enrollment
4. Pulmonary Arterial Hypertension not secondary to left heart disease
5. Contraindications to systemic anticoagulation
6. Hematocrit > 45%
7. Inability to obtain venous access
8. Hemodynamic instability severe enough to require IV positive inotropic agents, IV vasodilators or both
9. Use of iodinated radiocontrast material within the previous 72 hours or planned study requiring IV contrast during the current hospitalization
10. Severe concomitant disease expected to prolong hospitalization
11. Severe concomitant disease expected to cause death in ≤ 90 days
12. Sepsis or ongoing systemic infection
13. Severe uncorrected valvular stenosis
14. Active myocarditis
15. Hypertrophic obstructive cardiomyopathy
16. Constrictive pericarditis or restrictive cardiomyopathy
17. Liver cirrhosis
18. Previous solid organ transplant
19. Requirement for mechanical ventilatory support
20. Presence of a mechanical circulatory support device
21. Unwillingness or inability to complete follow up
22. Active drug or ETOH substance abuse
23. Participating in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosa Costanzo, MD, Principal Investigator — Midwest Heart Foundation
Locations (38):
- United States (38):
  - Heart Center Research, Huntsville, Alabama
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - Scottsdale Healthcare Research Institute, Scottsdale, Arizona
  - UCLA, Los Angeles, California
  - University of California, San Diego (UCSD), San Diego, California
  - San Diego Cardiac Center, San Diego, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Medical Center, Clearwater, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - Edward Hospital Center for Advanced Heart Failure, Naperville, Illinois
  - Advocate Health & Hospitals Corporation, Oakbrook Terrace, Illinois
  - Elkhart General HealthCare, Elkhart, Indiana
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - Iowa Health - Des Moines, Des Moines, Iowa
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Luke's Hospital and Saint Luke's Cardiovascular Consultants, Kansas City, Missouri
  - AtlantiCare Health Network, Egg Harbor, New Jersey
  - New Mexico Heart Institute/Heart Hospital, Albuquerque, New Mexico
  - Asheville Cardiology Associates, Asheville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Systems, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Oklahoma Heart Institute and Hillcrest Medical Center, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - St. Luke's Hospital and Health Network, Bethlehem, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Saint Thomas Hospital, Nashville, Tennessee
  - Brooke Army Medical Center, San Antonio, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - MultiCare Health System/Tacoma General Hospital, Tacoma, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Background] Costanzo MR, Guglin ME, Saltzberg MT, Jessup ML, Bart BA, Teerlink JR, Jaski BE, Fang JC, Feller ED, Haas GJ, Anderson AS, Schollmeyer MP, Sobotka PA; UNLOAD Trial Investigators. Ultrafiltration versus intravenous diuretics for patients hospitalized for acute decompensated heart failure. J Am Coll Cardiol. 2007 Feb 13;49(6):675-83. doi: 10.1016/j.jacc.2006.07.073. Epub 2007 Jan 26. PMID 17291932
- [Background] Adams KF Jr, Fonarow GC, Emerman CL, LeJemtel TH, Costanzo MR, Abraham WT, Berkowitz RL, Galvao M, Horton DP; ADHERE Scientific Advisory Committee and Investigators. Characteristics and outcomes of patients hospitalized for heart failure in the United States: rationale, design, and preliminary observations from the first 100,000 cases in the Acute Decompensated Heart Failure National Registry (ADHERE). Am Heart J. 2005 Feb;149(2):209-16. doi: 10.1016/j.ahj.2004.08.005. PMID 15846257
- [Background] Jain P, Massie BM, Gattis WA, Klein L, Gheorghiade M. Current medical treatment for the exacerbation of chronic heart failure resulting in hospitalization. Am Heart J. 2003 Feb;145(2 Suppl):S3-17. doi: 10.1067/mhj.2003.149. No abstract available. PMID 12594447
- [Background] Drazner MH, Rame JE, Stevenson LW, Dries DL. Prognostic importance of elevated jugular venous pressure and a third heart sound in patients with heart failure. N Engl J Med. 2001 Aug 23;345(8):574-81. doi: 10.1056/NEJMoa010641. PMID 11529211
- [Background] Domanski M, Norman J, Pitt B, Haigney M, Hanlon S, Peyster E; Studies of Left Ventricular Dysfunction. Diuretic use, progressive heart failure, and death in patients in the Studies Of Left Ventricular Dysfunction (SOLVD). J Am Coll Cardiol. 2003 Aug 20;42(4):705-8. doi: 10.1016/s0735-1097(03)00765-4. PMID 12932605
- [Background] Sharma A, Hermann DD, Mehta RL. Clinical benefit and approach of ultrafiltration in acute heart failure. Cardiology. 2001;96(3-4):144-54. doi: 10.1159/000047398. PMID 11805381
- [Background] Marenzi G, Lauri G, Grazi M, Assanelli E, Campodonico J, Agostoni P. Circulatory response to fluid overload removal by extracorporeal ultrafiltration in refractory congestive heart failure. J Am Coll Cardiol. 2001 Oct;38(4):963-8. doi: 10.1016/s0735-1097(01)01479-6. PMID 11583865
- [Background] Rimondini A, Cipolla CM, Della Bella P, Grazi S, Sisillo E, Susini G, Guazzi MD. Hemofiltration as short-term treatment for refractory congestive heart failure. Am J Med. 1987 Jul;83(1):43-8. doi: 10.1016/0002-9343(87)90495-5. PMID 3605181
- [Background] Jaski BE, Ha J, Denys BG, Lamba S, Trupp RJ, Abraham WT. Peripherally inserted veno-venous ultrafiltration for rapid treatment of volume overloaded patients. J Card Fail. 2003 Jun;9(3):227-31. doi: 10.1054/jcaf.2003.28. PMID 12815573
- [Background] Bart BA, Boyle A, Bank AJ, Anand I, Olivari MT, Kraemer M, Mackedanz S, Sobotka PA, Schollmeyer M, Goldsmith SR. Ultrafiltration versus usual care for hospitalized patients with heart failure: the Relief for Acutely Fluid-Overloaded Patients With Decompensated Congestive Heart Failure (RAPID-CHF) trial. J Am Coll Cardiol. 2005 Dec 6;46(11):2043-6. doi: 10.1016/j.jacc.2005.05.098. Epub 2005 Nov 4. PMID 16325039
- [Background] Costanzo MR, Saltzberg M, O'Sullivan J, Sobotka P. Early ultrafiltration in patients with decompensated heart failure and diuretic resistance. J Am Coll Cardiol. 2005 Dec 6;46(11):2047-51. doi: 10.1016/j.jacc.2005.05.099. Epub 2005 Nov 9. PMID 16325040
- [Background] Bart BA, Goldsmith SR, Lee KL, Givertz MM, O'Connor CM, Bull DA, Redfield MM, Deswal A, Rouleau JL, LeWinter MM, Ofili EO, Stevenson LW, Semigran MJ, Felker GM, Chen HH, Hernandez AF, Anstrom KJ, McNulty SE, Velazquez EJ, Ibarra JC, Mascette AM, Braunwald E; Heart Failure Clinical Research Network. Ultrafiltration in decompensated heart failure with cardiorenal syndrome. N Engl J Med. 2012 Dec 13;367(24):2296-304. doi: 10.1056/NEJMoa1210357. Epub 2012 Nov 6. PMID 23131078

RESULTS

PARTICIPANT FLOW:
Groups:
- Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration: Excess fluid from the patient was removed by isolated veno-venous ultrafiltration treatment using the FDA cleared Aquadex Flex Flow System during index hospitalization until the patient's signs and symptoms of fluid overload improved to the satisfaction of the treating physician. Diuretics were withheld for the duration of the AQ treatment and the use of positive inotropic agents and vasodilators were prohibited unless deemed necessary by the treating physician as rescue therapy. Ultrafiltration rates and monitoring of treatment were outlined in treatment guidelines.
- IV Loop Diuretics (LD): Excess fluid from the patient was removed by IV (Intravenous) loop diuretic treatment using only FDA approved IV loop diuretics indicated for the treatment of patients with fluid overload during index hospitalization until the patient's signs and symptoms of fluid overload improved to the satisfaction of the treating physician. This included furosemide or other IV loop diuretics administered at equivalent doses to furosemide. The recommended doses of IV bolus, maintenance dose and potential additional diuretics were outlined in treatment guidelines and were based on the CARRESS-HF Stepped Pharmacologic Protocol.
Period: Overall Study
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Started | 110 | 114
Completed | 81 | 84
Not Completed | 29 | 30

BASELINE CHARACTERISTICS:
Population: 3 patients in the IV Loop Diuretics (LD) arm were randomized, but withdrawn from the study prior to beginning study treatment. These patients are excluded from the number of baseline participants (analysis population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD) | Total
Number analyzed (Participants) | 110 | 111 | 221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.03 (12.61) | 66.87 (13.45) | 66.95 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 64
  Male | 76 | 81 | 157
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 30 | 61
  White | 75 | 71 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Height [Mean (Standard Deviation); unit: Centimeters] | 172.45 (11.04) | 174.12 (10.52) | 173.29 (10.79)
Weight [Mean (Standard Deviation); unit: Kilograms] | 110.06 (32.26) | 110.92 (35.09) | 110.49 (33.64)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 36.89 (10.13) | 36.32 (10.10) | 36.61 (10.10)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Heart Failure (HF) Event
Description: Time to first HF event within 90 days after discharge from index HF hospitalization. HF events are defined as
  * HF rehospitalization or
  * unscheduled outpatient or emergency room treatment with IV loop diuretics or
  * unscheduled outpatient Aquapheresis treatment
Time Frame: 90 days after discharge from index HF hospitalization.
Population: Results reported are for the 25th percentile.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 110 | 111
Days | 62 [42 to NA] — We are unable to estimate the upper limit of the confidence interval due to lack of events. | 34 [20 to 62]

2. Secondary Outcome: EFFICACY: Total Fluid Removed During the Index Hospitalization
Description: AQ-Fluid removed by AQ plus urine voided versus urine voided when treated with IV diuretics
Time Frame: Index Hospitalization, an average of 8 days
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 108 | 109
mL | 18700 (23033) | 14043 (15299)

3. Secondary Outcome: EFFICACY: Net Fluid Removed During the Index Hospitalization
Description: AQ-Fluid removed by AQ plus urine voided minus fluid intake versus urine voided minus fluid intake with the IV diuretics.
Time Frame: Index Hospitalization, an average of 8 days
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 108 | 109
mL | 12921 (20564) | 8907 (13329)

4. Secondary Outcome: EFFICACY: Weight Loss at 72 Hours After Initiation of Treatment
Description: Weight at 72 hours after treatment initiation minus weight at treatment initiation. Negative mean values indicate weight loss.
Time Frame: 72 hours after treatment initiation
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 85 | 82
lbs | -10.69 (7.20) | -10.30 (9.22)

5. Secondary Outcome: EFFICACY: Total Weight Loss During the Index Hospitalization
Description: Weight at hospital discharge minus weight at hospital admission. Negative mean values indicate weight loss.
Time Frame: Index Hospitalization, an average of 8 days
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 104 | 108
lbs | -17.12 (12.59) | -16.21 (14.23)

6. Secondary Outcome: EFFICACY: Time to Freedom From Congestion
Description: Time from hospital admission to time patient is free of congestion in the hospital. Freedom from congestion is defined as jugular venous distention of < or equal to 8 cm, with no orthopnea and with trace peripheral edema or no edema. Measurement taken every 24 hours after treatment initiation.
Time Frame: Index Hospitalization, an average of 8 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 40 | 46
Days | 5.28 (4.11) | 3.86 (3.23)

7. Secondary Outcome: EFFICACY: Freedom From Congestion
Description: Defined as jugular venous distention of < or equal to 8 cm, with no orthopnea, and with trace peripheral edema or no edema at hospital discharge
Time Frame: Index Hospitalization, an average of 8 days
Measure: Number; unit: Participants
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 110 | 111
Participants | 40 | 46

8. Secondary Outcome: EFFICACY: Changes in B-type Natriuretic Peptide (BNP) Levels Over Time
Description: Change in BNP levels over time at 72 hours, discharge, and 90 days after discharge.
Time Frame: Baseline and at 72 hours from baseline, hospital discharge and at 90 days after hospital discharge
Population: Number of participants analyzed changes over time. Baseline: n=108 for AQ arm, n=109 for LD arm. 72 hours from baseline: n=81 for AQ arm, n=77 for LD arm. Discharge: n=83 for AQ arm, n=89 for LD arm. 90 days follow up: n=65 for AQ arm, n=76 for LD arm.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 108 | 109
pg/mL
  Baseline | 814.0 (827.66) | 904.1 (843.44)
  72 hours from baseline | -169.8 (450.57) | -120.5 (469.04)
  Discharge | -250.2 (527.12) | -219.1 (539.26)
  90 days after discharge | -159.9 (678.20) | -201.3 (618.31)

9. Secondary Outcome: Length of Stay (LOS) During the Index Hospitalization
Description: Number of days patient is in hospital for HF treatment.
Time Frame: Index hospitalization admission to index hospitalization discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 105 | 108
Days | 8.49 (5.73) | 7.19 (5.37)

10. Secondary Outcome: CLINICAL: Total Number of Days Rehospitalized for Heart Failure (HF) at 30 and 90 Days After Discharge
Description: Days rehospitalized for HF symptoms requiring hospital, emergency room or clinic treatment involving the use of IV diuretics and /or positive inotropic or vasodilator drugs.
Time Frame: Within 30 days and 90 days after hospital discharge
Measure: Number; unit: Days
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 110 | 111
Days
  30 days after discharge | 68 | 172
  90 days after discharge | 338 | 460

11. Secondary Outcome: CLINICAL: Total Number of Emergency Department (ED) or Unscheduled Office Visits at 30 and 90 Days After Discharge
Description: Number of visits for HF symptoms requiring ED or clinic treatment involving the use of IV diuretics and /or positive inotropic or vasodilator drugs
Time Frame: Within 30 days and 90 days after hospital discharge
Measure: Number; unit: Visits
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 110 | 111
Visits
  30 days after discharge | 4 | 5
  90 days after discharge | 7 | 8

12. Secondary Outcome: CLINICAL: Total Number of Heart Failure (HF) Rehospitalizations at 30 and 90 Days After Discharge
Description: Number of different times patient was admitted to hospital for HF symptoms within 90 days of index hospitalization discharge.
Time Frame: Within 30 days and 90 days after hospital discharge
Measure: Number; unit: Rehospitalizations
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 110 | 111
Rehospitalizations
  30 days after discharge | 11 | 24
  90 days after discharge | 36 | 52

13. Secondary Outcome: CLINICAL: Total Number of Cardiovascular (CV) Rehospitalizations at 30 and 90 Days After Discharge
Description: CV symptoms that required hospitalization for treatment within 90 days of index hospitalization discharge.
Time Frame: Within 30 days and 90 days after hospital discharge
Measure: Number; unit: Rehospitalizations
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 110 | 111
Rehospitalizations
  30 days after discharge | 17 | 33
  90 days after discharge | 46 | 66

14. Secondary Outcome: CLINICAL: Total Number of Days for Cardiovascular (CV) Rehospitalizations at 30 and 90 Days After Discharge
Description: The total number of days spent in the hospital due to CV related events at 30 days and 90 days from hospital discharge.
Time Frame: Within 30 days and 90 days after hospital discharge
Measure: Number; unit: Days
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 110 | 111
Days
  30 days after discharge | 88 | 207
  90 days after discharge | 377 | 554

15. Secondary Outcome: CLINICAL: All Cause Rehospitalization Rates at 30 and 90 Days
Description: Any cause that required hospitalization for treatment within 90 days of index hospitalization discharge.
Time Frame: Within 30 days and 90 days after hospital discharge
Measure: Number; unit: Rehospitalizations/100 Pt-Days at Risk
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 110 | 111
Rehospitalizations/100 Pt-Days at Risk
  30 days after discharge | 0.899 | 1.278
  90 days after discharge | 1.109 | 1.237

16. Secondary Outcome: Mortality Rates Within Index Hospitalization or Within 90 Days After Hospital Discharge.
Description: Death due to any cause within index hospitalization and 90 days following hospital discharge.
Time Frame: Time from randomization to 90 days post-hospital discharge
Measure: Number; unit: Percentage of Participants
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 110 | 111
Percentage of Participants | 15.45 | 12.61

17. Secondary Outcome: Days Alive and Out of Hospital at 30 and 90 Days After Discharge
Description: Number of days patients were alive and out of the hospital at 30 and 90 days after discharge.
Time Frame: Within 30 and 90 days after hospital discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 105 | 108
Days
  30 days after discharge | 27.29 (5.78) | 26.46 (6.34)
  90 days after discharge | 62 (24.57) | 61.38 (24.95)

18. Secondary Outcome: Quality of Life Assessed Using the Kansas City Cardiomyopathy Questionnaire (KCCQ) at 30, 60 and 90 Days After Discharge
Description: Questionnaire assessed patients quality of life prior to index treatment versus timeframes following hospital discharge. Scores were transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Within 90 days after hospital discharge
Population: Number of participants analyzed changes over time. Baseline: n=107 for AQ arm, n=110 for LD arm. 30 day follow up: n=85 for AQ arm, n=91 for LD arm. 90 day follow up: n=72 for AQ arm, n=77 for LD arm.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 107 | 110
Scores on a Scale
  Baseline | 25.39 (19.37) | 28.64 (22.59)
  30 days after discharge | 52.06 (28.58) | 49.36 (28.82)
  90 days after discharge | 59.72 (24.90) | 58.50 (26.72)

19. Secondary Outcome: CLINICAL: Global Clinical Score at 30 and 90 Days After Discharge
Description: KCCQ Questionnaire analysis based on patient's self-assessment of how they feel at various intervals compared to how they felt prior to index treatment. Scores were transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Within 90 days after hospital discharge
Population: Number of participants analyzed changes over time. Baseline: n=107 for AQ arm, n=110 for LD arm. 30 day follow up: n=85 for AQ arm, n=92 for LD arm. 90 day follow up: n=72 for AQ arm, n=77 for LD arm.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 107 | 110
Scores on a Scale
  Baseline | 28.26 (18.65) | 31.83 (18.63)
  30 days after discharge | 54.78 (24.15) | 53.08 (26.01)
  90 days after discharge | 57.21 (25.39) | 60.56 (26.34)

20. Secondary Outcome: SAFETY: Changes in Renal Function (Serum Creatinine) After Treatment up to 90 Days After Randomization
Description: Changes in renal function prior to index treatment compared to various intervals by assessing the patient's serum creatinine (sCr), Blood Urea Nitrogen(BUN), BUN/sCr ratio and estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease (MDRD) formula
Time Frame: Within 90 days of randomization
Population: Number of participants analyzed changes over time. Discharge: n=105 for AQ arm, n=108 for LD arm. 30 days after discharge: n=93 for AQ arm, n=95 for LD arm. 60 days after discharge: n=85 for AQ arm, n=84 for LD arm. 90 days after discharge: n=4 for AQ arm, n=6 for LD arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 105 | 108
mg/dL
  Discharge | 0.12 (0.42) | 0.12 (0.50)
  30 days after discharge | 0.37 (3.41) | 0.17 (0.63)
  60 days after discharge | 1.34 (11.40) | -0.01 (0.44)
  90 days after discharge | -0.30 (0.42) | -0.24 (0.30)

21. Secondary Outcome: SAFETY: Changes in Renal Function (Blood Urea Nitrogen) After Treatment up to 90 Days After Randomization
Description: as for outcome 20
Time Frame: Within 90 days of randomization
Population: Number of participants analyzed changes over time. Baseline: n=105 for AQ arm, n=108 for LD arm. 30 days after discharge: n=93 for AQ arm, n=95 for LD arm. 60 days after discharge: n=85 for AQ arm, n=84 for LD arm. 90 days after discharge: n=4 for AQ arm, n=6 for LD arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 105 | 108
mg/dL
  Discharge | 8.38 (13.94) | 7.62 (14.34)
  30 days after discharge | 1.72 (14.44) | 6.56 (22.80)
  60 days after discharge | 1.85 (16.62) | 3.16 (17.78)
  90 days after discharge | 2.50 (6.36) | -3.78 (4.19)

22. Secondary Outcome: SAFETY: Changes in Renal Function (Blood Urea Nitrogen/Serum Creatinine) After Treatment up to 90 Days After Randomization
Description: as for outcome 20
Time Frame: Within 90 days of randomization
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 105 | 108
mg/dL
  Discharge | 3.77 (7.80) | 3.03 (6.52)
  30 days after discharge | 0.28 (6.88) | 1.65 (8.85)
  60 days after discharge | 0.07 (7.07) | 1.97 (7.42)
  90 days after discharge | 5.66 (1.40) | 1.72 (5.56)

23. Secondary Outcome: SAFETY: Changes in Renal Function (Estimated Glomerular Filtration Rate) After Treatment up to 90 Days After Randomization
Description: as for outcome 20
Time Frame: Within 90 days of randomization
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Number analyzed (Participants) | 105 | 108
mL/min/1.73m2
  Discharge | -2.31 (14.50) | -2.68 (13.45)
  30 days after discharge | -0.56 (14.24) | -3.33 (14.97)
  60 days after discharge | -2.49 (16.81) | 2.15 (13.79)
  90 days after discharge | 5.70 (8.06) | 7.41 (11.87)

ADVERSE EVENTS:
Time Frame: Baseline through 90 days after discharge.
Arm/Group | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration | IV Loop Diuretics (LD)
Serious Adverse Events (participants affected / at risk) | 73/110 | 67/111
Other Adverse Events (participants affected / at risk) | 25/110 | 18/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration (N=110) | IV Loop Diuretics (LD) (N=111)
Cardiac Failure (Cardiac disorders) | 5 | 8
Cardiac Failure Acute (Cardiac disorders) | 13 | 19
Cardiac Failure Congestive (Cardiac disorders) | 11 | 20
Chest Pain (General disorders) | 4 | 1
Pneumonia (Infections and infestations) | 5 | 0
Blood Creatinine Increase (Investigations) | 4 | 0
Renal Failure Acute (Renal and urinary disorders) | 4 | 3
Hypotension (Vascular disorders) | 3 | 5
Acute Coronary Syndrom (Cardiac disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 3 | 2
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 3 | 2
Cardiac Failure Chronic (Cardiac disorders) | 2 | 3
Cardio-Respiratory Arrest (Cardiac disorders) | 2 | 1
Cardiogenic Shock (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1
Cardiorenal Syndrome (Cardiac disorders) | 0 | 1
Cardiovascular Insufficiency (Cardiac disorders) | 1 | 0
Congestive Cardiomyopathy (Cardiac disorders) | 1 | 0
Cor Pulmonale (Cardiac disorders) | 0 | 2
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Right Ventricular Failure (Cardiac disorders) | 0 | 1
Supra Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 2 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Abdominal Wall Haematoma (Gastrointestinal disorders) | 1 | 0
Gastric Antral Vascular Ectasia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Cardiac Death (General disorders) | 0 | 1
Chest Discomfort (General disorders) | 1 | 0
Death (General disorders) | 0 | 3
Device Lead Issue (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Medical Device Complication (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Gallbladder Perforation (Hepatobiliary disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 2
Filariasis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic Shock (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Renal Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular Graft Thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Anticoagulation Drug Level Below Therapeautic (Investigations) | 1 | 0
Cardiac Output Decreased (Investigations) | 1 | 0
Haematocrit Decreased (Investigations) | 1 | 0
International Normalised Ratio Increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Cerebrovascular Disorder (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Neurological Symptom (Nervous system disorders) | 2 | 1
Neuropathy Peripheral (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Failure Chronic (Renal and urinary disorders) | 2 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac Ablation (Surgical and medical procedures) | 0 | 1
Cardioversion (Surgical and medical procedures) | 1 | 2
Implantable Defibrillator Insertion (Surgical and medical procedures) | 3 | 0
Ventricular Assist Device Insertion (Surgical and medical procedures) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aquapheresis (AQ) - Isolated Veno-venous Ultrafiltration (N=110) | IV Loop Diuretics (LD) (N=111)
Blood Creatinine Increase (Investigations) | 7 | 4
Hypotension (Vascular disorders) | 12 | 7
Urinary Tract Infection (Infections and infestations) | 3 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 4
Renal Failure Acute (Renal and urinary disorders) | 5 | 7

LIMITATIONS AND CAVEATS:
Due to patient recruitment challenges, the study was terminated early. At that time, no interim analyses of the data had been completed; therefore the decision to close the study was not related to any underlying concerns about safety or futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other